CLINICAL TRIAL: NCT02025842
Title: Long-term Nucleoside/Nucleotide Treatment of Hepatitis B Virus HBeAg-negative Genotype D Patients and Risk of Hepatocellular Carcinoma:Evidence From the CLEO Cohort Study
Brief Title: Hepatitis B Virus HBeAg-negative Genotype D Patients and Hepatocellular Carcinoma
Acronym: HBV/HCC
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Responsible Party: Principal Investigator, Adriano Pellicelli, medical doctor, Azienda Ospedaliera San Camillo Forlanini
Other Study IDs: 02
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Hepatocellular Carcinoma; Hepatitis B
Keywords: Hepatocellular carcinoma; Hepatitis B
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 62 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chronic hepatitis B patients: Chronic hepatitis B patients treated with nucleoside/nucleotide
- Compensated cirrhosis patients: Compensated cirrhosis patients treated with nucleoside/nucleotide

SUMMARY:
To evaluate the impact of liver fibrosis and other variables [e.g., age, sex, virological response (VR), and previous resistance to nucleoside/nucleotide analogue (NUC) therapy] on Hepatocellular carcinoma incidence in an Italian population of genotype D HBeAg-negative CHB patients treated with long-term NUC therapy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) usually develops in patients with chronic liver disease, particularly patients with liver cirrhosis. Chronic hepatitis B (CHB) is one of the most frequent underlying causes of HCC. Several studies have demonstrated that variations in the hepatitis B virus (HBV) genotype have different effects on HCC. HBV genotypes C and D had lower responses to interferon-based therapy and higher frequencies of basal core promoter mutations than genotypes A and B.For this reason, HBV genotypes C and D seem to lead to more severe liver disease, including cirrhosis, compared with the other HBV genotypes. Because liver cirrhosis is one of the strongest HCC risk factors in CHB patients, antiviral therapy may prevent the development of liver complications such as HCC. The aim of this study is to evaluate the impact of liver fibrosis and other variables, such as age, sex, virological response (VR), and resistance to nucleoside/nucleotide analogue (NUC) therapy, in a population of genotype D HBeAg-negative CHB patients treated with long-term NUC therapy.

ELIGIBILITY:
Inclusion Criteria:

* Only chronic hepatitis B or compensated cirrhosis HBeAg-negative genotype D patients were included in this study.The patients were included in this study if they were ≥18 years old and had received treatment with nucleoside/nucleotide for a period of at least 18 months.

Exclusion Criteria:

* Patients with Hepatocellular carcinoma diagnosed before or during the first 18 months of nucleoside/nucleotide therapy, as well as patients coinfected with hepatitis D, hepatitis C, or HIV, were excluded. Patients with decompensated cirrhosis were excluded because of the low number of cases observed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2000 to December 2013, 745 HBV-infected patients were included in the database. Of these, 438 were excluded: 226 did not fulfil the diagnosis of CHB, 75 had HBeAg-positive CHB, 20 had received NUC for <18 months, 26 had HCC diagnosed before or within the first 18 months of therapy, and 61 presented a different HBV genotype. Thirty patients had decompensated cirrhosis. A total of 306 HBeAg-negative genotype D patients were selected and included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2000-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
risk for hepatocellular carcinoma | follow-up of 62.5 months (range, 18 to 112 months),
  The primary endpoint of the study was the development of Hepatocellular carcinoma. We assessed the risk of development of hepatocellular carcinoma according to liver status, viral response to treatment, and the presence of previous resistance to NUC therapy.

SECONDARY OUTCOMES:
survival | follow-up of 62.5 months (range, 18 to 112 months),
  survival in cirrhosis and chronic hepatitis B patients

CONTACTS AND LOCATIONS:
Overall Officials: Adriano M Pellicelli, MD, Principal Investigator — AO San Camillo Forlanini